CLINICAL TRIAL: NCT06116955
Title: The Application of Balanced Propofol Sedation in Fiberoptic Bronchoscopy
Status: Completed | Type: Observational
Sponsor: The Affiliated Hospital of Qingdao University (Other)
Responsible Party: Principal Investigator, jixiangyu, Principal Investigator, The Affiliated Hospital of Qingdao University
Other Study IDs: QYFYEC2023-111
Record Dates: First submitted 2023-10-25; First posted 2023-11-03 (Actual); Last update posted 2024-01-31 (Actual); Status verified 2024-01

CONDITIONS: Bronchoscopy
Keywords: Propofol; Balanced propofol sedation; Remazolam; Bronchoscopy
MeSH Terms: interventions — Midazolam; Sufentanil; Propofol

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- S-M group: Midazolam combines with sufentanil to titrate to moderate sedation for bronchoscopy.
  Interventions: Drug: Midazolam and sufentanil
- S-M-P group: Midazolam and sufentanil combine with low-dose propofol to titrate to deep sedation for bronchoscopy.
  Interventions: Drug: Midazolam, sufentanil and propofol
- S-R group: Remazolam combines with sufentanil to titrate to moderate sedation for bronchoscopy.
  Interventions: Drug: Remazolam and sufentanil.
- S-R-P group: Remazolam and sufentanil combine with low-dose propofol to titrate to deep sedation for bronchoscopy.
  Interventions: Drug: Remazolam, sufentanil and propofol

INTERVENTIONS:
Drug: Midazolam and sufentanil — Patients undergoing bronchoscopic diagnosis and treatment under moderate sedation with midazolam combined with sufentani.
  Groups: S-M group
Drug: Midazolam, sufentanil and propofol — Patients undergoing bronchoscopic diagnosis and treatment under deep sedation with midazolam and sufentani combined with propofol.
  Groups: S-M-P group
Drug: Remazolam and sufentanil. — Patients undergoing bronchoscopic diagnosis and treatment under moderate sedation with remazolam combined with sufentani.
  Groups: S-R group
Drug: Remazolam, sufentanil and propofol — Patients undergoing bronchoscopic diagnosis and treatment under deep sedation with remazolam and sufentani combined with propofol.
  Groups: S-R-P group

SUMMARY:
The purpose of this study is to investigate the feasibility of using balanced propofol sedation for bronchoscopy. And screen out the optimal balanced propofol sedation compatibility plan.

DETAILED DESCRIPTION:
Balanced propofol sedation (BPS) is a technique proposed and developed by gastroenterologists. In recent years, multiple studies have confirmed that the use of BPS in gastrointestinal endoscopy can not only ensure patient comfort, but also reduce the incidence of respiratory and circulatory suppression. Moreover, the postoperative recovery time is short. Even for non-anesthesiologists applying BPS in gastrointestinal endoscopy , it has high safety.

Compared with gastrointestinal endoscopy, bronchoscopy occupies the respiratory tract and most patients have respiratory system diseases. Therefore, it is more necessary for strict respiratory management and control of patient sedation depth. Traditional midazolam combined with opioid drugs or propofol monosedation cannot effectively meet clinical needs. The excellent sedative and analgesic effects of BPS, as well as its maintenance of respiratory and circulatory functions, make it theoretically very suitable for application in bronchoscopy. However, there is currently a lack of evidence to support the application of BPS in bronchoscopy.

ELIGIBILITY:
Inclusion Criteria:

1. American Society of Anesthesiologists classes I-IV ;
2. Patients undergo painless bronchoscopy, including bronchoscopic biopsy (bronchoscopic lesion biopsy, bronchial mucosal biopsy, bronchoscopic transmural lung biopsy, bronchoscopic needle aspiration biopsy) ,bronchoalveolar lavage and bronchoscopic treatment;
3. Normal communication skills and able to cooperate in completing this study;
4. Patients who voluntarily accept this experimental study and sign the "Trial Informed Consent Form".

Exclusion Criteria:

1. Patients with contraindications or allergies to anesthesia;
2. Individuals with a history of alcoholism or drug abuse;
3. Patients with contraindications for puncture of the cricoid membrane;
4. Patients with mental or neurological disorders, taking anti anxiety/depression drugs, or primary diseases with laboratory evidence indicating possible changes in hormone levels;
5. Patients with difficulty in language communication, poor understanding ability, and inability to cooperate in completing experimental studies;
6. Patients who require laryngeal mask or tracheal intubation for assisted ventilation during the examination process;
7. Patients undergoing rigid bronchoscopy treatment;
8. Patients who refuse to receive sedation or have not signed the "Trial Informed Consent Form".

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Population undergoing bronchoscopy examination at Qingdao University Affiliated Hospital from December 2023 to January 2014.
Sampling Method: Non-Probability Sample
Enrollment: 424 (Actual)
Dates: Start 2023-09-21 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2024-01-01 (Actual)

PRIMARY OUTCOMES:
Patient satisfaction | During bronchoscopy.
  The investigator needs to use VAS scores to evaluate satisfaction about sedation feeling when they accepted bronchoscopy. The score from 0 (extremely dissatisfied) to 10 (extremely satisfied).
Clinical satisfaction | During bronchoscopy.
  The investigator needs to use VAS scores to evaluate satisfaction about doctors and nurses when they carry out the operation. The score from 0 (extremely dissatisfied) to 10 (extremely satisfied).
Patient's recovery time | The end of bronchoscopy (up to 2 hours).
  The investigator needs to record the wake-up time of patients after the end of bronchoscopy.
Patient's departure time | The end of bronchoscopy (up to 2 hours).
  The investigator needs to record the patient's departure time after the end of bronchoscopy.

SECONDARY OUTCOMES:
Induction time | Before bronchoscopy.
  Time from administering sedative and analgesic drugs to titration with propofol until MOAA/S 2-3 points.
Drug dosage | Before bronchoscopy and during bronchoscopy.
  Induced, maintenance and total dose of midazolam, propofol.
Additional frequency of propofol during bronchoscopy | During bronchoscopy.
  Additional frequency of propofol during bronchoscopy.
Additional frequency of 2% lidocaine during bronchoscopy | During bronchoscopy.
  Additional frequency of 2% lidocaine during bronchoscopy.
Additional dosage of 2% lidocaine during bronchoscopy | During bronchoscopy.
  Additional dosage of 2% lidocaine during bronchoscopy.
Additional dosage of propofol during bronchoscopy | During bronchoscopy.
  Additional dosage of propofol during bronchoscopy.
Patient response score during bronchoscopy | During bronchoscopy.
  Researcher used the Behavioral Pain Scale for non intubated patients (BPS-NI) to assess their response scores. The tool consists of 3 behavioral domains: facial expressions, movements, and vocalization. The total BPS-IN value can range from 3 (no pain) to 12 (most pain).
Adverse reactions during bronchoscopy | During bronchoscopy
  Record the number of occurrences of hypotension, hypertension, tachycardia, bradycardia, arrhythmias, hypoxemia, apnea, coughing (no wheezing during continuous coughing, considered as one coughing), and physical activity (non directive limb activity) during bronchoscopy.
  After fully awake, researcher 2 used the VAS score for adverse reactions during the resuscitation process, such as dizziness, pain, nausea, breathing difficulties, etc.
Adverse reactions after fully awake | The end of bronchoscopy (up to 2 hours).
  After fully awake, researcher used the VAS score for adverse reactions during the resuscitation process, such as dizziness, pain, nausea, breathing difficulties, etc. The score from 0 (no uncomfortable) to 10 (extremely uncomfortable).
Patient's anxiety/depression state | Day before bronchoscopy. 1, 3, 7, and 14 days after bronchoscopy.
  Researcher used the Patient Health Questionnaire-8 (PHQ-8) to assess Patient's anxiety/depression state. The total score range of PHQ-8 is 0-24. No depressive symptoms on a score of 0-4, mild on a score of 5-9, moderate on a score of 10-14, and severe on a score of 15 or above.

CONTACTS AND LOCATIONS:
Locations (1):
- Affiliated Hospital of Qingdao University, Shandong, Qingdao, China